CLINICAL TRIAL: NCT06306261
Title: Controlling the Mental Health for a Better Response to Treatment in Patients With Ulcerative Colitis
Acronym: TIMAEUS
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Professore, IRCCS San Raffaele
Other Study IDs: TIMAEUS
Record Dates: First submitted 2024-02-20; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients in remission of the disease: UC patients will be subjected to a questionnaire every month about their habits.
  Interventions: Other: questionnaire
- patients in reactivation of the disease: UC patients will be subjected to a questionnaire every month about their habits.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — UC patients will be subjected to a questionnaire each month about their habits.

SUMMARY:
The project aims to implement the Internet Of Thing (IoT) platform of the San Raffaele Hospital (OSR) with data from stress conditions perceived by the patient through the synergistic collaboration between patients, gastroenterologists and psychologists.

DETAILED DESCRIPTION:
This is a prospective, single-center observational study involving patients with an established diagnosis of UC who are currently receiving standard care and eligible for advanced therapies at the San Raffaele Hospital (OSR).

The estimated sample size for the 1-year project is 150 UC patients eligible for advanced therapy.

This study aims to understand the relationship between environmental factors, dietary composition, and altered intestinal permeability that contribute to flares in UC patients by leveraging Internet-Of-Things (IoT) technologies.

These subjects will be asked to answer a series of questions about feelings and thoughts via the mobile app each month.

The mobile app was developed and designed following the open source ResearchKit framework.

The questionnaire based on the Perceived Stress Scale (PSS) will be created thanks to the collaboration between the gastroenterologist and psychologists of the San Raffaele Hospital (OSR). The PSS is a classic stress assessment tool.

Finally, all this data will be integrated thanks to the bioinformatic tool based on machine learning. All analyzes will be performed and stored in a dedicated cloud service (https://www.heroku.com/), which will make the project feasible and easy to manage.

ELIGIBILITY:
Inclusion Criteria:

- Patients in whom the ulcerative colitis has been diagnosed and eligible for advanced therapies Patients will be asked to sign an informed consensus before filling out the questionnaire.

Exclusion Criteria:

- Patients in whom the ulcerative colitis has not been diagnosed. All those who have not signed previously informed consensus.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 patients affected by UC under the standard of care protocols at OSR, will be subjected to a questionnaire each 30 days about their habits.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
to evaluate mental stress/health as an impacting factor on UC progression | 8 months
  The enrolled UC patients should compile a questionnaire which asks about feelings and thoughts.
  The questionnaire will be the Italian version of the Perceived Stress Scale (PSS).
  The scale goes from 0 to 4.Scoring is reversed for positive questions 0= 4 scores; 1= 3 scores, 2=2 scores; 3=1 score; 4=0. For negative questions are 0 minimum score and 4 maximum score Higher score is considered more stress, so worse outcome, conversely lower score is less stress so better outcome.
  Patients will be remembered to answer to questions about their habits though a notification every 30 days in mobile app.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Ospedale San Raffaele, Milan, Italy